CLINICAL TRIAL: NCT04741269
Title: Asymmetric Lack of Knee Flexion as a Symptom of DLM in Children
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1241
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Highlights a New Clinical Sign Which Point Out a Meniscus Posterior Luxation Because of a MCA-type DLM
Keywords: discoid lateral meniscus; children; instability; arthroscopy; repair; lack of flexion; flexion block knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lack of knee flexion: During preoperative clinical exam, highlight of a lack of knee flexion. The lack of knee flexion consists in an asymmetric heel-bottom distance or an asymmetric goniometric measure of knee flexion.
  All others characteristics are also analyzed like in group 2, as : rest of knee motion, MRI meniscus shift, arthroscopic shift
  Interventions: Diagnostic Test: Find a link between lack of knee flexion and meniscal posterior luxation fixed
- Full knee flexion: During preoperative clinical exam, highlight of a lack of knee flexion. The lack of knee flexion consists in an asymmetric heel-bottom distance or an asymmetric goniometric measure of knee flexion. Patients in group 2 don't have any asymmetric full knee flexion.
  All others characteristics are also analyzed like in group 2, as : rest of knee motion, MRI meniscus shift, arthroscopic shift

INTERVENTIONS:
Diagnostic Test: Find a link between lack of knee flexion and meniscal posterior luxation fixed — Measure the full flexion angle of the knee using a goniometer. Measure the heel-buttom distance. All measurements are carried out in bilateral and comparative ways.
  Search for the meniscal position on MRI and intraoperatively: no shift, anterior, medial, posterior shift.
  Groups: Lack of knee flexion

SUMMARY:
Highlighted during the clinical examination of a knee flexion asymmetry, and related to the intraoperative meniscal observations on DLM.

Search for a link between asymmetric bending defect and posterior shift in MCA-type DLM.

Analysis of all patients with symptomatic DLM.

ELIGIBILITY:
Inclusion Criteria:

* < 18 yo
* Symptomatic discoid lateral meniscus

Exclusion Criteria:

* Osteochondritis dissecans (OCD)
* Asymptomatic and partial DLM observed during arthroscopic exploration for other reasons
* Revision knee surgery

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with a discoid lateral meniscus symptomatic and surgical care.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Meniscal posterior shift per-operative | During surgery for MCA-type DLM
  Visualization of a dislocated posterior meniscus during arthroscopy, before any reduction or meniscoplasty procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas CANCE, MD, Principal Investigator — Paediatric orthopaedic - Femme Mère Enfant Hospital (HFME)
Locations (1):
- Paediatric orthopaedic - Femme Mère Enfant Hospital (HFME), Lyon, France